CLINICAL TRIAL: NCT02980289
Title: DAnish Nausea Study In Advanced Cancer-Epidemiology: A Danish Multicenter Trial to Investigate the Prevalence and Treatment of Nausea and/or Vomiting in Patients With Advanced Cancer.
Status: Completed | Type: Observational
Sponsor: Signe Harder (Other)
Responsible Party: Sponsor-Investigator, Signe Harder, Doctor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: DANSAC-EPI
Record Dates: First submitted 2016-03-07; First posted 2016-12-02 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Advanced Cancer; Nausea; Emesis
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients over 18 years old with advanced cancer defined as metastatic disease, no curable treatment options. The patients may not have received chemotherapy or irradiation within 4 weeks, no operations within 2 weeks and no general anesthesia within 4 days.

SUMMARY:
The study aims to investigate the prevalence and treatment of nausea and/or vomiting in patients with advanced cancer not receiving chemotherapy or irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced cancer
2. Age ≥ 18 years
3. Ability to read and understand the forms required for the study
4. Life-expectancy more than 2 weeks.
5. Nausea score ≥ 'a little' on the extended EORTC QLQ-C15-PAL (item 9)

Exclusion Criteria:

1. Surgery to the brain or abdomen within the last 2 weeks or exposure to general anesthesia within the last 4 days.
2. Chemotherapy or radiation therapy within the last 4 weeks
3. Symptoms of increased intracranial pressure or cerebral metastasis. If this is suspected, a normal MRI scan of the cerebrum is needed before inclusion
4. Radiologically confirmed ileus, or strong clinical suspicion evaluated by the study Investigator
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer, who have not received chemo- or radiotherapy in the last 4 weeks prior to screening, will be screened for nausea and/or vomiting following evaluation of the primary inclusion-/exclusion criteria. The patients can be located either in the hospital departments, at home or in a hospice.
Sampling Method: Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
2-item nausea-score from EORTC-QLQ-C15-Pal at baseline and 1 week | From baseline and at 1 week (5-9 days)
  The primary objective is to observe the effect of standard anti-emetics on change in two-item nausea-score from baseline to 24 hours.

SECONDARY OUTCOMES:
Nausea CAT-score from EORTC-QLQ-C15-Pal at baseline and after 1 week | 1 week (5-9 days)
  Change in nausea CAT-score from baseline to 24 hours and 7 days
Nausea at screening from EORTC-QLQ-C15-Pal at baseline | At baseline
  Prevalence of nausea at time of screening, related to age, cancer-diagnosis and gender
Emesis at screening from EORTC-QLQ-C15-Pal at baseline | At baseline
  Prevalence of emesis at time of screening, related to age, cancer-diagnosis and gender
Change in other parameters from EORTC-QLQ-C15-Pal at baseline and after 1 week | From baseline and at 1 week (5-9 days)
  Change in other parameters potentially indicative of efficacy: appetite, fatigue, pain, emotional function and overall quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Odense Universityhospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No